CLINICAL TRIAL: NCT01368133
Title: The Observational Study of the Structures and Functions of Multiple Organs in Patients With Growth Hormone-secreting Tumors
Brief Title: The Observational Study of Growth Hormone-secreting Pituitary Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Zhaoyun Zhang, Associate Professor, Huashan Hospital
Other Study IDs: 2010M-010
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Acromegaly; Pituitary Tumor
Keywords: acromegaly; pituitary tumor
MeSH Terms: conditions — Acromegaly; Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, DNA and pituitary tumor tissues
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The major purpose of this study is to evaluate the changes of multiple organs in patients with growth hormone-secreting pituitary tumors before and after surgery. Plasma, DNA samples and pituitary tumor tissues will be kept for further analysis.

DETAILED DESCRIPTION:
Multiple organs or systems will be affected by excessive growth hormones in patients with acromegaly. The major purpose of this study is to evaluate the changes before and after the pituitary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acromegaly
* > 18 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The acromegaly patients at Huashan Hospital will be recruited anf followed up prior to surgery and one month, 3 months, 6 months and 12 months after surgery.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhao, M.D., Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China